CLINICAL TRIAL: NCT03000036
Title: Doxorubicin-associated Cardiac Tissue Remodeling Followed by CMR of Myocardial Extracellular Volume and Myocyte Size in Breast Cancer Patients
Brief Title: Doxorubicin-associated Cardiac Remodeling Followed by CMR in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Otavio Rizzi Coelho Filho, Professor, University of Campinas, Brazil
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DOX-0675014600011
Record Dates: First submitted 2016-11-28; First posted 2016-12-21 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer Female; Doxorubicin Induced Cardiomyopathy
Keywords: Breast cancer; Doxorubicin; Cardiovascular Magnetic Resonance; T1 mapping
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; gadoterate meglumine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiovascular Magnetic Resonance (Other): Twenty-seven female patients were imaged in a 3T magnet after consecutively enrolled in the study if they had received a breast cancer diagnosis at the Center for Integral Attention to Women's Health (University of Campinas) and had prescribed endovenous doxorubicin as part of their chemotherapy regimen.
  Interventions: Drug: Doxorubicin; Device: Achieva, Philips Medical Systems (3T magnet); Drug: Gadoterate Meglumine

INTERVENTIONS:
Drug: Doxorubicin — Patients had prescribed endovenous doxorubicin as part of their chemotherapy regimen (mean cumulative dose 102,66 mg/m2, administered in 4 doses with 21 days interval).
  Other Names: Adriamycin
Device: Achieva, Philips Medical Systems (3T magnet) — Patients were imaged in supine position in a 3T magnet (Achieva, Philips Medical Systems, Best, The Netherlands). The protocol consisted of electrocardiographically gated cine imaging with steady state free-precession to assess left ventricular (LV) ejection fraction and LV mass. For imaging of late gadolinium-DTPA enhancement (LGE) we used an inversion-recovery-prepared, gradient-echo sequence with segmented acquisition, which was triggered every other heartbeat. LGE images were acquired during end-expiratory breath-holding, after administration of Dotarem. T1 was performed with a Look-Locker sequence with a non-slice-selective adiabatic inversion pulse, followed by segmented gradient-echo acquisition for 17 times after inversion, covering approximately two cardiac cycles. T1 imaging was repeated in the same LV short-axis slice, once before and five to seven times after the injection of gadolinium to cover an approximately 30-min period of slow contrast clearance.
  Other Names: Cardiovascular Magnetic Resonance (CMR)
Drug: Gadoterate Meglumine — LGE images were acquired starting within 10 min after bolus administration of a cumulative dose of 0.2 mmol/Kg of gadoterate meglumine (Dotarem, Guerbet, Aulnay-sous-Bois, France).
  Other Names: Dotarem

SUMMARY:
Twenty-seven breast cancer women without heart failure, underwent CMR imaging (3T-Achieva, Philips) before and 3 times serially after 4-cycles of adjuvant DOX (60mg/m2). CMR assessed left ventricular (LV) ejection fraction (EF), T1 mapping pre and post gadolinium and late gadolinium enhancement imaging. Biomarkers were obtained before and 72 hours after each DOX-cycle.

DETAILED DESCRIPTION:
This prospective cohort study was performed at the State University of Campinas, Brazil. The Institutional Review Board of the State University of Campinas approved the study and all participants provided informed consent. Female patients with breast cancer who received anthracycline (doxorubicin or daunorubicin or epirubicin) as part of their chemotherapy protocol were enrolled in the study.

Detailed medical history, standard anthropometric data, and measurement hemogram, troponin, CKMB, cholesterol, serum glucose, CRP and biomarkers were obtained.

As in adults, chronic anthracycline-related cardiotoxicity typically presents early, within one year after termination of chemotherapy and the peak time for the appearance of symptoms of heart failure is about three months after the last anthracycline dose, patients underwent CMR before and three times serially after DOX (two, five and twelve months).

Patients were imaged in supine position in a 3T magnet (Achieva, Philips Medical Systems, Best, The Netherlands). The CMR protocol consisted of electrocardiographically gated cine imaging with steady state free-precession to assess left ventricular (LV) function and LV mass. For imaging of late gadolinium enhancement (LGE) we used an inversion-recovery-prepared, gradient-echo sequence with segmented acquisition, which was triggered every other heartbeat. LGE images were acquired during end-expiratory breath-holding for slices matching the slice locations for cine imaging, starting within 10 min after bolus administration of a cumulative dose of 0.2 mmol/Kg of gadoterate meglumine (Dotarem, Guerbet, Aulnay-sous-Bois, France). T1 was performed with a Look-Locker sequence with a non-slice-selective adiabatic inversion pulse, followed by segmented gradient-echo acquisition for 17 times after inversion, covering approximately two cardiac cycles. The Look-Locker sequence was performed in a single short-axis slice at the level of the mid left ventricle. T1 imaging was repeated in the same LV short-axis slice, once before and five to seven times after the injection of gadolinium to cover an approximately 30-min period of slow contrast clearance.

All images were analyzed with MASS CMR software (Mass Research, Leiden University Medical Center, Leiden, the Netherlands). For LV mass and function quantification, the endocardial and epicardial borders of the LV myocardium were manually traced on short-axis cine images at end-diastole and systole. Papillary muscles were excluded from LV mass, and LV mass was indexed to body surface area.

For each Look-Locker image series, the endocardial and epicardial borders of the LV were traced and divided into six standard segments. Signal intensity versus time curves for each segment and the blood pool were used to determine segmental T1* by nonlinear, least-squares fitting to an analytic expression for the magnitude signal measured during the inversion recovery. T1 was calculated from the T1* and the amplitude parameters to correct for the effects of radiofrequency pulses applied during the inversion recovery.

Pairs of R1 values for myocardial tissue and blood data were fit with a two-space water-exchange model of equilibrium transcytolemmal water exchange. The myocardial extracellular volume fraction (ECV) and the intracellular lifetime of water (τic), a cell size-dependent parameter, were adjustable parameters of this model. The measured blood hematocrit was a fixed parameter of the model. All R1 measurements for each patient were used to fit the model to determine ECV and τic.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer and had prescribed an anthracycline agent as part of their chemotherapy regimen

Exclusion Criteria:

* Strict contraindications to MRI
* Acute or chronic kidney failure
* Previously diagnosed myocardial infarction, heart failure, valvular disease or cardiomyopathy.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-07; Primary Completion 2015-01 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Quantification of fibrosis index by Cardiac Magnetic Resonance | two years
  Estimate the extracellular volume fraction derived from gadolinium-DTPA partition Coefficient of the myocardium
Intracellular lifetime of water (τic) by Cardiac Magnetic Resonance | two years
  This metric estimates the myocyte size using Cardiac Magnetic Resonance T1 mapping data

SECONDARY OUTCOMES:
Left ventricular mass by Cardiac Magnetic Resonance | two years
  Electrocardiographically gated cine imaging with steady state free-precession to assess left ventricular mass.
Left ventricular volumes by Cardiac Magnetic Resonance | two years
  Electrocardiographically gated cine imaging with steady state free-precession to assess left ventricular volume.
Left ventricular ejection fraction by Cardiac Magnetic Resonance | two years
  Electrocardiographically gated cine imaging with steady state free-precession to assess left ventricular ejection fraction.
Left ventricular myocardial edema fraction by Cardiac Magnetic Resonance | two years
  Using T2-weighted sequences to visualize myocardial edema

OTHER OUTCOMES:
Ultra-sensitive troponin | two years
  Cardiac troponin (ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Otávio R. Coelho-Filho, MD, MPH, PhD, Principal Investigator — University of Campinas, Brazil
Locations (1):
- State University of Campinas, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim RJ, Wu E, Rafael A, Chen EL, Parker MA, Simonetti O, Klocke FJ, Bonow RO, Judd RM. The use of contrast-enhanced magnetic resonance imaging to identify reversible myocardial dysfunction. N Engl J Med. 2000 Nov 16;343(20):1445-53. doi: 10.1056/NEJM200011163432003. PMID 11078769
- [Background] Kim RJ, Fieno DS, Parrish TB, Harris K, Chen EL, Simonetti O, Bundy J, Finn JP, Klocke FJ, Judd RM. Relationship of MRI delayed contrast enhancement to irreversible injury, infarct age, and contractile function. Circulation. 1999 Nov 9;100(19):1992-2002. doi: 10.1161/01.cir.100.19.1992. PMID 10556226
- [Background] Tandri H, Saranathan M, Rodriguez ER, Martinez C, Bomma C, Nasir K, Rosen B, Lima JA, Calkins H, Bluemke DA. Noninvasive detection of myocardial fibrosis in arrhythmogenic right ventricular cardiomyopathy using delayed-enhancement magnetic resonance imaging. J Am Coll Cardiol. 2005 Jan 4;45(1):98-103. doi: 10.1016/j.jacc.2004.09.053. PMID 15629382
- [Background] Hunold P, Wieneke H, Bruder O, Krueger U, Schlosser T, Erbel R, Barkhausen J. Late enhancement: a new feature in MRI of arrhythmogenic right ventricular cardiomyopathy? J Cardiovasc Magn Reson. 2005;7(4):649-55. doi: 10.1081/jcmr-65608. PMID 16136854
- [Background] Harris PA, Lorenz CH, Holburn GE, Overholser KA. Regional measurement of the Gd-DTPA tissue partition coefficient in canine myocardium. Magn Reson Med. 1997 Oct;38(4):541-5. doi: 10.1002/mrm.1910380406. PMID 9324319
- [Background] Flacke SJ, Fischer SE, Lorenz CH. Measurement of the gadopentetate dimeglumine partition coefficient in human myocardium in vivo: normal distribution and elevation in acute and chronic infarction. Radiology. 2001 Mar;218(3):703-10. doi: 10.1148/radiology.218.3.r01fe18703. PMID 11230643
- [Background] Elliott P. Pathogenesis of cardiotoxicity induced by anthracyclines. Semin Oncol. 2006 Jun;33(3 Suppl 8):S2-7. doi: 10.1053/j.seminoncol.2006.04.020. PMID 16781283
- [Background] Iles L, Pfluger H, Phrommintikul A, Cherayath J, Aksit P, Gupta SN, Kaye DM, Taylor AJ. Evaluation of diffuse myocardial fibrosis in heart failure with cardiac magnetic resonance contrast-enhanced T1 mapping. J Am Coll Cardiol. 2008 Nov 4;52(19):1574-80. doi: 10.1016/j.jacc.2008.06.049. PMID 19007595
- [Background] Ellinor PT, Sasse-Klaassen S, Probst S, Gerull B, Shin JT, Toeppel A, Heuser A, Michely B, Yoerger DM, Song BS, Pilz B, Krings G, Coplin B, Lange PE, Dec GW, Hennies HC, Thierfelder L, MacRae CA. A novel locus for dilated cardiomyopathy, diffuse myocardial fibrosis, and sudden death on chromosome 10q25-26. J Am Coll Cardiol. 2006 Jul 4;48(1):106-11. doi: 10.1016/j.jacc.2006.01.079. Epub 2006 Jun 21. PMID 16814656
- [Background] Ong DS, Scherrer-Crosbie M, Coelho-Filho O, Francis SA, Neilan TG. Imaging methods for detection of chemotherapy-associated cardiotoxicity and dysfunction. Expert Rev Cardiovasc Ther. 2014 Apr;12(4):487-97. doi: 10.1586/14779072.2014.893824. PMID 24650314
- [Background] Kehr E, Sono M, Chugh SS, Jerosch-Herold M. Gadolinium-enhanced magnetic resonance imaging for detection and quantification of fibrosis in human myocardium in vitro. Int J Cardiovasc Imaging. 2008 Jan;24(1):61-8. doi: 10.1007/s10554-007-9223-y. Epub 2007 Apr 12. PMID 17429755
- [Background] Flett AS, Hayward MP, Ashworth MT, Hansen MS, Taylor AM, Elliott PM, McGregor C, Moon JC. Equilibrium contrast cardiovascular magnetic resonance for the measurement of diffuse myocardial fibrosis: preliminary validation in humans. Circulation. 2010 Jul 13;122(2):138-44. doi: 10.1161/CIRCULATIONAHA.109.930636. Epub 2010 Jun 28. PMID 20585010
- [Background] Swain SM. Doxorubicin-induced cardiomyopathy. N Engl J Med. 1999 Feb 25;340(8):654; author reply 655. No abstract available. PMID 10049087
- [Background] Aiken MJ, Suhag V, Garcia CA, Acio E, Moreau S, Priebat DA, Chennupati SP, Van Nostrand D. Doxorubicin-induced cardiac toxicity and cardiac rest gated blood pool imaging. Clin Nucl Med. 2009 Nov;34(11):762-7. doi: 10.1097/RLU.0b013e3181b7d76f. PMID 19851170
- [Background] Ewer MS, O'Shaughnessy JA. Cardiac toxicity of trastuzumab-related regimens in HER2-overexpressing breast cancer. Clin Breast Cancer. 2007 Jun;7(8):600-7. PMID 17592672
- [Background] Perez EA. Cardiac toxicity of ErbB2-targeted therapies: what do we know? Clin Breast Cancer. 2008 Mar;8 Suppl 3:S114-20. doi: 10.3816/cbc.2008.s.007. PMID 18777950
- [Background] Chien AJ, Rugo HS. The cardiac safety of trastuzumab in the treatment of breast cancer. Expert Opin Drug Saf. 2010 Mar;9(2):335-46. doi: 10.1517/14740331003627441. PMID 20175700
- [Background] Cardinale D, Sandri MT, Colombo A, Colombo N, Boeri M, Lamantia G, Civelli M, Peccatori F, Martinelli G, Fiorentini C, Cipolla CM. Prognostic value of troponin I in cardiac risk stratification of cancer patients undergoing high-dose chemotherapy. Circulation. 2004 Jun 8;109(22):2749-54. doi: 10.1161/01.CIR.0000130926.51766.CC. Epub 2004 May 17. PMID 15148277
- [Background] Ewer MS, Lenihan DJ. Left ventricular ejection fraction and cardiotoxicity: is our ear really to the ground? J Clin Oncol. 2008 Mar 10;26(8):1201-3. doi: 10.1200/JCO.2007.14.8742. Epub 2008 Jan 28. No abstract available. PMID 18227525
- [Background] Von Hoff DD, Rozencweig M, Layard M, Slavik M, Muggia FM. Daunomycin-induced cardiotoxicity in children and adults. A review of 110 cases. Am J Med. 1977 Feb;62(2):200-8. doi: 10.1016/0002-9343(77)90315-1. PMID 835599
- [Background] Von Hoff DD, Layard MW, Basa P, Davis HL Jr, Von Hoff AL, Rozencweig M, Muggia FM. Risk factors for doxorubicin-induced congestive heart failure. Ann Intern Med. 1979 Nov;91(5):710-7. doi: 10.7326/0003-4819-91-5-710. PMID 496103
- [Background] Coelho-Filho OR, Mongeon FP, Mitchell R, Moreno H Jr, Nadruz W Jr, Kwong R, Jerosch-Herold M. Role of transcytolemmal water-exchange in magnetic resonance measurements of diffuse myocardial fibrosis in hypertensive heart disease. Circ Cardiovasc Imaging. 2013 Jan 1;6(1):134-41. doi: 10.1161/CIRCIMAGING.112.979815. Epub 2012 Nov 15. PMID 23159497
- [Background] Rickers C, Wilke NM, Jerosch-Herold M, Casey SA, Panse P, Panse N, Weil J, Zenovich AG, Maron BJ. Utility of cardiac magnetic resonance imaging in the diagnosis of hypertrophic cardiomyopathy. Circulation. 2005 Aug 9;112(6):855-61. doi: 10.1161/CIRCULATIONAHA.104.507723. PMID 16087809
- [Background] Landis CS, Li X, Telang FW, Molina PE, Palyka I, Vetek G, Springer CS Jr. Equilibrium transcytolemmal water-exchange kinetics in skeletal muscle in vivo. Magn Reson Med. 1999 Sep;42(3):467-78. doi: 10.1002/(sici)1522-2594(199909)42:33.0.co;2-0. PMID 10467291
- [Background] Coelho-Filho OR, Shah RV, Mitchell R, Neilan TG, Moreno H Jr, Simonson B, Kwong R, Rosenzweig A, Das S, Jerosch-Herold M. Quantification of cardiomyocyte hypertrophy by cardiac magnetic resonance: implications for early cardiac remodeling. Circulation. 2013 Sep 10;128(11):1225-33. doi: 10.1161/CIRCULATIONAHA.112.000438. Epub 2013 Aug 2. PMID 23912910
- [Derived] Ferreira de Souza T, Quinaglia A C Silva T, Osorio Costa F, Shah R, Neilan TG, Velloso L, Nadruz W, Brenelli F, Sposito AC, Matos-Souza JR, Cendes F, Coelho OR, Jerosch-Herold M, Coelho-Filho OR. Anthracycline Therapy Is Associated With Cardiomyocyte Atrophy and Preclinical Manifestations of Heart Disease. JACC Cardiovasc Imaging. 2018 Aug;11(8):1045-1055. doi: 10.1016/j.jcmg.2018.05.012. PMID 30092965